CLINICAL TRIAL: NCT06985524
Title: Clinical and Preparation Studies of Traditional Chinese Medicine Compound(Weipi Formula) in the Treatment of Epigastric Stuffiness Syndrome
Brief Title: To Observe the Clinical Efficacy of Traditional Chinese Medicine Compound(Weipi Formula ) in the Treatment of Epigastric Stuffiness Syndrome
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240108120356554
Record Dates: First submitted 2025-05-14; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Functional Dyspepsia(FD) Was Studied

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Weipi Formula (Experimental): Participants will take Weipi Formula（Wu SiSi Formula）for 2 weeks.
  Interventions: Drug: Weipi Formula（Wu SiSi Formula）
- Arm placebo (Experimental)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Weipi Formula（Wu SiSi Formula） — take Weipi Formula（Wu SiSi Formula） or the placebo daily for 2 weeks.
  Arms: Arm Weipi Formula
Other: Placebo — Take Weipi Formula（Wu SiSi Formula） or the placebo daily for 2 weeks.
  Arms: Arm placebo

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy of the herbal drug Weipi formula in treating functional dyspepsia (FD) in adults. It will also assess the safety of Weipi formula. The main questions the study aims to answer are:

Does Weipi formula reduce participants' TCM syndrome scores? What medical issues might participants experience while taking Weipi formula?

Researchers will compare Weipi formula with a placebo (an identical-looking substance without active drugs) to determine whether Weipi formula is effective in treating functional dyspepsia.

Participant Procedures

Participants will:

Take Weipi formula or the placebo daily for 2 weeks.

Visit the clinic once every week for examinations and tests. Record their symptoms and undergo measurements (e.g., pepsin levels).

ELIGIBILITY:
Inclusion Criteria:

* ① Meet the diagnostic criteria for epigastric fullness (Pi-Man) in Traditional Chinese Medicine (TCM);

  * Meet the Western diagnostic criteria for functional dyspepsia (FD), specifically postprandial distress syndrome (PDS) subtype, or meet both PDS and epigastric pain syndrome (EPS) subtypes but with PDS as the dominant presentation;

    * Age 18-80 years;

      * Willing to sign the informed consent form.

Exclusion Criteria:

* ① Gastroscopy findings: Benign or malignant digestive diseases (e.g., peptic ulcer, gastric cancer);

  * Severe organic diseases of the liver, gallbladder, spleen, or pancreas;

    * Severe organic diseases in other organ systems;

      * Pregnant or lactating women; ⑤ Patients with psychiatric disorders causing similar symptoms (e.g., schizophrenia, anxiety disorder, major depressive disorder); ⑥ Regular use (≥3 months) of NSAIDs and/or selective COX-2 inhibitors; ⑦ Potassium supplements taken within 2 weeks prior to enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
TCM syndrome scores | From enrollment to the end of treatment at 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- he Second Affiliated Hospital of Nanchang University, No. 1 Minde Road, Donghu District, Nanchang City, Jiangxi Province, China, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No